CLINICAL TRIAL: NCT03475628
Title: A Prospective, Multicenter, Non-comparative, Open-label, Phase II Study to Evaluate the Effects of Daratumumab Monotherapy on Bone Parameters in Patients With Relapsed and /or Refractory Multiple Myeloma Who Have Received at Least 2 Prior Lines of Therapy, Including Lenalidomide and a Proteasome Inhibitor
Brief Title: Effects of Daratumumab Monotherapy on Bone Parameters in Patients With Relapsed and /or Refractory Multiple Myeloma
Acronym: REBUILD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hellenic Society of Hematology (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EAE-2017/MM01
Record Dates: First submitted 2018-02-22; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Intervention Model Description: Single arm: Daratumumab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daratumumab (Experimental): Daratumumab at a dose of 16 mg/kg administered as an IV infusion at weekly intervals (QW) for 8 weeks, then every 2 weeks (Q2W) for an additional 16 weeks, then every 4 weeks (Q4W) thereafter.
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Daratumumab will be given at a dose of 16 mg/kg administered as an IV infusion at weekly intervals (QW) for 8 weeks, then every 2 weeks (Q2W) for an additional 16 weeks, then every 4 weeks (Q4W) thereafter. Subjects will receive pre-infusion medications prior to Daratumumab infusion to mitigate potential IRRs and post- infusion medications after Daratumumab infusion for the prevention of delayed IRRs

SUMMARY:
The purpose of this study is to evaluate the effects of daratumumab monotherapy on bone disease in patients with relapsed/refractory MM who have received at least 2 prior lines of therapy, including lenalidomide and a PI.

DETAILED DESCRIPTION:
This is a prospective, multicenter, non-comparative, open-label Phase II study. Daratumumab will be administered according to approved label. Approximately 57 subjects located in Greece will be enrolled in the study.

Patients shall receive treatment until disease progression, physician decision, unacceptable toxicity, withdrawal of consent, or death (whichever occurs first). Survival status and data of subsequent anti-myeloma treatment will be collected post-treatment.

Primary and secondary variables related to bone disease markers will be evaluated every other cycle of therapy. Disease evaluations will occur monthly and consist mainly of measurements of myeloma proteins. Other parameters may include bone marrow examinations, skeletal surveys, assessment of extramedullary plasmacytomas, and measurements of serum calcium corrected for albumin, and β2- microglobulin and albumin. Assessment of myeloma response and disease progression will be conducted in accordance with the modified IMWG response criteria

ELIGIBILITY:
Inclusion Criteria:

1. Males and females at least 18 years of age.
2. Voluntary written informed consent.
3. Subject must have documented relapsed or refractory multiple myeloma as defined by the criteria below:

   a. Measurable disease as defined by any of the following:
   * Serum monoclonal paraprotein (M-protein) level ≥ 1.0 g/dL (except for IgA subtype: ≥ 0.5 g/dL) or urine M-protein level ≥ 200 mg/24 hours; or
   * Light chain multiple myeloma for subjects without measurable disease in the serum or urine by SPEP/UPEP: Serum immunoglobulin free light chain ≥ 10 mg/dL and abnormal serum immunoglobulin kappa lambda free-light-chain ratio.
4. Prior treatment with at least two lines of therapy including lenalidomide and a PI for MM (induction followed by any planned high dose therapy or consolidation or maintenance would be considered as one regimen).
5. Documented evidence of progressive disease as defined by the IMWG 2014 on or after the last regimen.
6. Karnofsky Performance Status score of ≥ 70.
7. All of the following laboratory test results during screening:

   * Absolute neutrophil count (ANC) of ≥1.0 x 109/L.
   * Platelet count of ≥ 75 x 109/L in patients in whom <50% of bone marrow nucleated cells are plasma cells and ≥50 x 109/L in patients in whom more than 50% of bone marrow nucleated cells are plasma cells.
   * Hemoglobin value (> 7.5 g/dL).
   * Alanine aminotransferase level ≤2.5 times the upper limit of normal (ULN).
8. Adequate renal function (CrCl ≥ 30 mL/min by CKD-EPI).
9. Willingness and ability to participate in study procedures.
10. Reproductive Status:

    1. Women of childbearing potential (WOCBP) must have two negative serum or urine pregnancy tests, one 10-14 days prior to start of the study drug and one within 24 hours prior to the start of study drug.
    2. Women must not be breastfeeding.
    3. WOCBP must agree to follow instructions for effective methods of contraception for 4 weeks before the start of treatment with study drugs, for the duration of treatment with study drugs, and for 3 months after cessation of study treatment.

Male patients must use a latex or synthetic condom during any sexual contact with females of reproductive potential, even if they have undergone a successful vasectomy. They must also agree to follow instructions for methods of contraception for 4 weeks before the start of treatment with study drugs, for the duration of treatment with study drugs, and for a total of 3 months post-treatment completion.

Exclusion Criteria:

1. Patient has received any of the following therapies:

   * Radiotherapy or systemic therapy within 2 weeks of baseline.
   * Prior Allogeneic hematopoietic stem cell transplantation within 12 weeks of baseline.
   * Prior Treatment with any CD38-antibody (i.e. isatuximab).
2. Clinically significant cardiac disease, including:

   1. Myocardial infarction within 6 months, or unstable or uncontrolled condition (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV).
   2. Cardiac arrhythmia (CTCAE Grade 3 or higher) or clinically significant ECG abnormalities.
   3. ECG showing a baseline QT interval as corrected >470 msec.
3. Chronic obstructive pulmonary disease (COPD) with a Forced Expiratory Volume in 1 second (FEV1) <50% of predicted normal. Note that FEV1 testing is required for subjects suspected of having COPD and subjects must be excluded if FEV1 <50% of predicted normal.
4. Known active hepatitis A, B, or C.
5. Known HIV infection.
6. Significant neuropathy (Grades 3-4, or Grade 2 with pain) within 14 days prior to enrolment.
7. Hypersensitivity to the active substance or to any of the excipients.
8. Any concurrent medical or psychiatric condition or disease (e.g., active systemic infection, uncontrolled diabetes, acute diffuse infiltrative pulmonary disease) that is likely to interfere with subject's ability to give informed consent, the study procedures or results, or that in the opinion of the investigator, would constitute a hazard for participating in this study.
9. Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2018-02-21 (Actual); Primary Completion 2019-06-20 (Estimated); Study Completion 2020-02-20 (Estimated)

PRIMARY OUTCOMES:
changes in bone resorption marker, C-telopeptide of collagen type 1 (CTX), after 4 months of daratumumab monotherapy | assessed on baseline and after 4 months from initiation of daratumumab monotherapy
  The evaluation of the changes in bone resorption marker after 4 months of daratumumab monotherapy. CTX (measured in pg/ml) will be evaluated at baseline and then every 2 months of therapy.
changes in bone resorption marker, namely, tartrate-resistant acid phosphatase-5b (TRACP-5b) after 4 months of daratumumab monotherapy | assessed on baseline and after 4 months from initiation of daratumumab monotherapy
  The evaluation of the changes in bone resorption marker after 4 months of daratumumab monotherapy. TRACP-5b (measured in mU/dL) will be evaluated at baseline and then every 2 months of therapy

SECONDARY OUTCOMES:
Changes in bone formation marker, bALP. | from baseline up to 12 months of daratumumab monotherapy or at end of treatment
  Change from baseline in bone formation marker bALP (measured in U/L) after 4, 8 and 12 months of daratumumab monotherapy (or at the end of therapy)
Changes in bone formation marker, OC. | from baseline up to 12 months of daratumumab monotherapy or at end of treatment
  Change from baseline in bone formation marker OC (measured in ng/ml) after 4, 8 and 12 months of daratumumab monotherapy (or at the end of therapy)
Changes in bone formation marker, PINP. | from baseline up to 12 months of daratumumab monotherapy or at end of treatment
  Change from baseline in bone formation marker PINP (measured in ng/ml) after 4, 8 and 12 months of daratumumab monotherapy (or at the end of therapy)
Changes in bone resorption marker, CTX. | from baseline up to12 months of daratumumab monotherapy or at end of treatment
  Change from baseline in bone resorption marker CTX (measured in pg/ml) after 8 and 12 months of daratumumab monotherapy
Changes in bone resorption marker, TRACP-5b. | from baseline up to12 months of daratumumab monotherapy or at end of treatment
  Change from baseline in bone resorption marker TRACP-5b (measured in mU/dL) after 8 and 12 months of daratumumab monotherapy
Changes in bone marker RANKL | from baseline up to 12 months of daratumumab monotherapy or at end of treatment
  Change from baseline in RANKL (measured in pg/ml) after 4, 8 and 12 months of daratumumab monotherapy
Changes in bone marker ratio,RANKL/OPG ratio. | from baseline up to 12 months of daratumumab monotherapy or at end of treatment
  Change from baseline in RANKL/OPG ratio after 4, 8 and 12 months of daratumumab monotherapy
Changes in bone marker CCL3 | from baseline up to 12 months of daratumumab monotherapy or at end of treatment
  Change from baseline in CCL3 (measured in pg/ml) after 4, 8 and 12 months of daratumumab monotherapy
Changes in bone marker Dkk1 | from baseline up to 12 months of daratumumab monotherapy or at end of treatment
  Change from baseline in Dkk1 (measured in ng/ml) after 4, 8 and 12 months of daratumumab monotherapy
Changes in bone marker SOST | from baseline up to 12 months of daratumumab monotherapy or at end of treatment
  Change from baseline in SOST (measured in pmol/L) after 4, 8 and 12 months of daratumumab monotherapy
Changes in bone marker activin-A | from baseline up to 12 months of daratumumab monotherapy or at end of treatment
  Change from baseline in activin-A (measured in μg/L) after 4, 8 and 12 months of daratumumab monotherapy
Change in Bone Mineral Density (BMD) of lumbar spine | measured at baseline and after 6 and 12 months after initiation of daratumumab monotherapy
  Change in Bone Mineral Density (BMD) of lumbar spine measured by DXA after 6 and 12 months of daratumumab monotherapy
Immunomodulatory effects of daratumumab on T cells by comprehensive molecular and phenotypic studies and correlations with bone markers | : measured at baseline and after 3 and 6 months after initiation of daratumumab monotherapy
  Immunomodulatory effects of daratumumab on T cells by comprehensive molecular and phenotypic studies and correlations with bone markers
Progression free survival (PFS) | from recruitment to the date of the first documented PD or death due to any cause, whichever comes first (approximately up to 2 years).
  Progression free survival is defined as the time, in months, from recruitment to the date of the first documented PD or death due to any cause, whichever comes first. PD will be assessed by the investigator based on the analysis of serum and urine protein electrophoresis (sPEP and uPEP), serum free light chain protein (sFLC), Corrected serum calcium assessment, imaging and bone marrow assessments as per modified IMWG guidelines.
Overall survival | Time from first dose of study treatment to death (approximately up to 2 years)
  Overall survival is defined as the time, in months
Time to next treatment | From first dose until the date to next anti-neoplastic therapy or death from any cause, whichever comes first (approximately up to 2 years)
  Time to next therapy will be defined as the time, in months.
Spinal cord compression (Skeletal surveys-Skeletal related events) | From baseline to 24 months (up to 2 years)
  Spinal cord compression will be evaluated in terms of number (and percentage) of patients with events and number of events per patient
The incidence of pathological fractures (Skeletal surveys-Skeletal related events) | From baseline to 24 months (up to 2 years)
  The incidence of pathological fractures will be evaluated in terms of number (and percentage) of patients with events and number of events per patient
Need for radiotherapy or surgery to the bones (Skeletal surveys-Skeletal related events) | From baseline to 24 months (up to 2 years)
  Need for radiotherapy or surgery to the bones will be evaluated in terms of number (and percentage) of patients with events and number of events per patient
Safety (adverse events) | Continuously throughout the study, starting from informed consent until 30 days after last study treatment (approximately up to 30 months)
  The incidence of Adverse Events will be assessed according to the common Terminology Criteria for Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Terpos, Assoc Prof, Principal Investigator — Department of Clinical therapeutics, National and Kapodistrian University of Athens, School of medicine, Athens, Greece
Locations (1):
- General Hospital of Athens "Alexandra", Athens, Attica, Greece